CLINICAL TRIAL: NCT06197984
Title: Exploring Antimicrobial Resistance in Patients With Acute Cholangitis Undergoing ERCP: A Prospective Multicentre Study
Brief Title: Antimicrobial Resistance in Acute Cholangitis
Acronym: ARISE
Status: Recruiting | Type: Observational
Sponsor: Emergency County Hospital Pius Brinzeu; Timisoara, Romania (Network)
Collaborators: Carol Davila University of Medicine and Pharmacy (Other); Grigore T. Popa University of Medicine and Pharmacy (Other); Bucharest Emergency Hospital (Other)
Responsible Party: Principal Investigator, Bogdan Miutescu, MD, MD,PhD, Emergency County Hospital Pius Brinzeu; Timisoara, Romania
Other Study IDs: 407/29.09.2023
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cholangitis Acute; Biliary Tract Diseases; Jaundice; Malignant; Jaundice, Obstructive; Choledocholithiasis
Keywords: Acute Cholangitis; Antibiotics; MultiDrug Resistance (MDR)
MeSH Terms: conditions — Biliary Tract Diseases; Jaundice; Jaundice, Obstructive; Choledocholithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute cholangitis: Patients admitted to the hospital due to acute cholangitis and undergoing ERCP will be selected. Bile specimens will be obtained after cannulation through the sphincterotome before the therapeutic intervention.
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — ERCP will serve as the exclusive therapeutic modality, aided by a therapeutic duodenoscope to access the common bile duct using a guidewire.

SUMMARY:
This study prospectively explores antimicrobial resistance in patients with acute cholangitis undergoing ERCP procedures. By analyzing patient profiles, microbial cultures, and treatment outcomes, the current study seeks to identify specific patterns of resistance, assess the effectiveness of current antimicrobial therapies, and explore potential strategies to optimize treatment regimens.

DETAILED DESCRIPTION:
Given the extensive utilization of antibiotics and the worldwide rise of multidrug-resistant organisms, there are ongoing initiatives to ascertain microbiological traits and discern patterns of drug resistance associated with intra-abdominal infections.

Microbial cultures from bile and blood samples will be established and characterized using appropriate methodologies. For patients with moderate and severe acute cholangitis (AC), blood cultures will be initiated upon admission, adhering to the Tokyo Guidelines for AC 2018 recommendations. Bile specimens will be obtained after cannulation through the sphincterotome before the therapeutic intervention. Initially, a minimum of 5 mL of the procured bile will be discarded, followed by the collection of an additional 5 mL in a sterile vessel containing a medium conducive to both anaerobic and aerobic bacterial cultures. The samples will undergo a minimum incubation period of seven days at 37 °C until microbial proliferation becomes evident. Antibiotic susceptibility assessments, specifically minimum inhibitory concentration (MIC), will be performed and interpreted according to established guidelines.The analysis of samples will occur within the laboratory of each respective center, with antibiograms conducted in accordance with established protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute cholangitis
* Ability to provide an informed consent
* Age over 18 years
* Any gender

Exclusion Criteria:

* Age under 18
* Pregnancy
* Post-ERCP perforation
* The patient's decision to abstain from study enrollment
* Patients unable to express informed consent
* Patients from whom a bile sample could not be collected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital with acute cholangitis undergoing ERCP as part of routine medical care.
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Exploring antimicrobial resistance of bile cultures and characterizing bacterial profile | 2 years
  The primary objective of this prospective, multicenter study is to meticulously characterize the bacterial profile and assess the antimicrobial resistance of bile cultures in patients diagnosed with acute cholangitis undergoing ERCP procedures. By employing advanced microbiological analyses, the investigators aim to identify specific bacterial strains and their resistance profiles, providing comprehensive insights into the dynamics of infection. This primary outcome will contribute to the development of tailored antimicrobial strategies, optimizing the management and treatment outcomes for individuals with acute cholangitis.

SECONDARY OUTCOMES:
Isolated bacteria and the etiology of obstructive biliary disease | 2 years
  Secondary objectives encompass exploring the correlation between isolated bacteria and the etiology of obstructive biliary disease.
Multidrug-Resistance (MDR) | 2 years
  Additionally, the investigators aim to determine the occurrence and frequency of multidrug-resistant (MDR) organisms and sentinel microorganisms in bile samples.
ERCP naive patients vs. patients with a history of ERCP | 2 years
  Furthermore, the investigators are going to explore potential variations in the biliary microbial community, making comparisons between patients with no prior ERCP experience (naive) and those with a history of ERCP procedures. This comprehensive secondary outcome analysis seeks to unravel microbial relationships, antibiotic resistance patterns, and the impact of procedural history on biliary microbial communities in the context of acute cholangitis.

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Miutescu, MD,PhD, Principal Investigator — Emergency County Hospital Pius Brinzeu; Timisoara, Romania
Locations (1):
- Bogdan Miutescu, Timișoara, Romania

IPD SHARING:
Plan to Share IPD: No